CLINICAL TRIAL: NCT02717624
Title: A Phase 1b, Multicenter, Open-label Study of Acalabrutinib in Combination With Bendamustine and Rituximab (BR) or Venetoclax and Rituximab (VR) in Subjects With Mantle Cell Lymphoma
Brief Title: A Study of Acalabrutinib in Combination With Rituximab + (Bendamustine or Venetoclax) in Subjects With MCL
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Acerta Pharma BV (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACE-LY-106; 2023-509353-31-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2016-02-24; First posted 2016-03-24 (Estimated); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Mantle Cell Lymphoma (MCL)
Keywords: Bruton Tyrosine Kinase Inhibitor; BTK; Mantle Cell Lymphoma; MCL; Acalabrutinib; ACE-LY-106
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — acalabrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1: Acalabrutinib+BR in TN patients (Experimental): Part 1: Acalabrutinib in combination with drugs bendamustine and rituximab (BR) in treatment naive patients
  Interventions: Drug: Acalabrutinib in combination with BR
- Part 1: Acalabrutinib+BR in RR patients (Experimental): Part 1: Acalabrutinib in combination with bendamustine and rituximab (BR) in relapse refractory patients
  Interventions: Drug: Acalabrutinib in combination with BR
- Part 2: Acalabrutinib+VR in TN patients (Experimental): Part 2: Acalabrutinib in combination with venetoclax and rituximab (VR) in treatment naive patients
  Interventions: Drug: Acalabrutinib in combination with VR

INTERVENTIONS:
Drug: Acalabrutinib in combination with BR
  Other Names: Acalabrutinib + BR
  Arms: Part 1: Acalabrutinib+BR in RR patients; Part 1: Acalabrutinib+BR in TN patients
Drug: Acalabrutinib in combination with VR
  Other Names: Acalabrutinib + VR
  Arms: Part 2: Acalabrutinib+VR in TN patients

SUMMARY:
A Phase 1b, Multicenter, Open-label Study of Acalabrutinib in Combination with Bendamustine and Rituximab (BR) or Venetoclax and Rituximab (VR) in Subjects with Mantle Cell Lymphoma

DETAILED DESCRIPTION:
This is a multicenter, open-label Phase 1b study to assess the safety and efficacy of acalabrutinib when administered concomitantly with bendamustine and rituximab in subjects with treatment naive or relapse refractory mantle cell lymphoma (Part 1), or when administered concomitantly with venetoclax and rituximab in subjects with treatment naive mantle cell lymphoma (Part 2).

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥ 18 years of age.
* Pathologically confirmed MCL.
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2.
* Agreement to use highly effective forms of contraception during the study and for 2 days after the last dose of acalabrutinib, 30 days after the last dose of venetoclax, or 12 months after the last dose of rituximab, whichever is longest.
* Treatment Naive MCL patients requiring treatment with no exposure to prior therapies.

Exclusion Criteria:

* Significant cardiovascular disease such as uncontrolled or untreated symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening, or any Class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification.Exception: Subjects with controlled, asymptomatic atrial fibrillation during screening are allowed to enroll on study
* Malabsorption syndrome, disease significantly affecting gastrointestinal function, resection of the stomach, extensive small bowel resection that is likely to affect absorption, symptomatic inflammatory bowel disease, partial or complete bowel obstruction, or gastric restrictions and bariatric surgery, such as gastric bypass
* Uncontrolled active systemic fungal, bacterial, viral, or other infection (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment), or intravenous anti-infective treatment within 2 weeks before first dose of study drug
* Breastfeeding or pregnant
* Concurrent participation in another therapeutic clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2016-04-20 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2027-08-20 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment Emergent Adverse Events (AEs) as assessed by CTCAE v4.03 | From first dose of study drug to within 30 days of last dose of study drug
  Number of participants who had experienced at least one treatment emergent AE

CONTACTS AND LOCATIONS:
Overall Officials: Acerta Clinical Trials, Study Director — 1-888-292-9613; acertamc@dlss.com
Locations (14):
- United States (9):
  - Research Site, Louisville, Kentucky
  - Research Site, Ann Arbor, Michigan
  - Research Site, Hackensack, New Jersey
  - Research Site, Morristown, New Jersey
  - Research Site, Lake Success, New York
  - Research Site, Columbus, Ohio
  - Research Site, Nashville, Tennessee
  - Research Site, Houston, Texas
  - Research Site, Seattle, Washington
- Research Site, Bologna, Italy
- Poland (4):
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Olsztyn
  - Research Site, Warsaw

REFERENCES:
- [Derived] Wang M, Robak T, Maddocks KJ, Phillips T, Smith SD, Gallinson D, Calvo R, Wun CC, Munugalavadla V, Jurczak W. Acalabrutinib plus venetoclax and rituximab in treatment-naive mantle cell lymphoma: 2-year safety and efficacy analysis. Blood Adv. 2024 Sep 10;8(17):4539-4548. doi: 10.1182/bloodadvances.2023012424. PMID 38781315